CLINICAL TRIAL: NCT05152030
Title: Validation of the Local Applicability of the 'TIB' Olfactory Test Device in the Era of COVID-19
Brief Title: The Clinical Applicability of the 'TIB' Olfactory Test Device
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CE20329A#1
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Anosmia; Hyposmia
MeSH Terms: conditions — Anosmia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- hyposmic patients
  Interventions: Diagnostic Test: 'TIB' Olfactory Test; Diagnostic Test: Traditional Chinese version of the University of Pennsylvania of Smell Identification Test (UPSIT-TC)
- anosmic patients
  Interventions: Diagnostic Test: 'TIB' Olfactory Test; Diagnostic Test: Traditional Chinese version of the University of Pennsylvania of Smell Identification Test (UPSIT-TC)
- normosmic group
  Interventions: Diagnostic Test: 'TIB' Olfactory Test; Diagnostic Test: Traditional Chinese version of the University of Pennsylvania of Smell Identification Test (UPSIT-TC)

INTERVENTIONS:
Diagnostic Test: 'TIB' Olfactory Test — A new smell identification test, 'TIB' Olfactory Test Device (Top International Biotech, Taipei) has been developed in Taiwan. It consists of 16 tests with an odorant embedded in fragrant microcapsules positioned on a strip. The examinee scratches the strip to release the odorant. The released odorant is sniffed and the examinee identifies the odorant by choosing a name from a set of 4 odor descriptors. This process is then repeated with the next odorant on the strip.
Diagnostic Test: Traditional Chinese version of the University of Pennsylvania of Smell Identification Test (UPSIT-TC) — The University of Pennsylvania Smell Identification Test (UPSIT), which was developed at the University of Pennsylvania, is one of the most reliable and the most widely used olfactory test.The test consists of four 10-odorant booklets. Each odorant is embedded in 10 to 50 µm urea-formaldehyde polymer microencapsules fixed in a proprietary binder and positioned on a brown strip which is located at the bottom of each page of the test booklet.4 When the examinee takes the test, each of the 40 odorants is released by scratching the strip with a pencil tip. The released odorant is sniffed and the examinee identifies the odorant by choosing a name from a set of 4 odor descriptors.

SUMMARY:
The aim of this study was to evaluate the validity and test-retest reliability of the 'TIB' Olfactory Test Device, a new olfactory test tool developed by Top International Biotech, Taipei, and to determine its normative values. The olfactory function of 180 subjects was evaluated using both the traditional Chinese version of the University of Pennsylvania of Smell Identification Test (UPSIT-TC) and TIB. The subjects consisted of 60 healthy volunteers (normosmic group), 60 hyposmic patients, and 60 anosmic patients. The healthy volunteers were retested with the UPSIT-TC and TIB at an inter-test interval of at least 7 days. The cut-off scores of TIB among the different groups were determined by receiver operating characteristic curve.

ELIGIBILITY:
Inclusion Criteria:

* Normosmic group were self-reported absence of deficits in olfaction. Hyposmic patients were loss of olfactory function with a phenyl ethyl alcohol (PEA) odor detection threshold below -1. Anosmic patients were loss of olfactory function with a PEA threshold equal to -1.

Exclusion Criteria:

* History of sinonasal symptoms within a week before the test

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normosmic group were from community. Hyposmic and anosmic patients were from out patient clinic department of Otorhinolaryngology.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
validity of TIB olfactory test | 30 minutes to 1 hour
  Criterion validity: Correlation between UPSIT-TC and TIB olfactory test
Reliability of TIB olfactory test | 1 week
  Test-retest reliability

CONTACTS AND LOCATIONS:
Overall Officials: Rong-San Jiang, M.D., Ph.D., Study Director — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan